CLINICAL TRIAL: NCT03715309
Title: R2 in the Treatment of Follicular Lymphoma Grade 1-3A
Brief Title: R2 in the Treatment of Follicular Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-R2
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Revlimd (Experimental)
  Interventions: Drug: Revlimid

INTERVENTIONS:
Drug: Revlimid — Revlimid 25mg PO d1-10 Plus Rituximab 375 mg/m2 IV d0
  Other Names: lenalidomide

SUMMARY:
Lenalidomide Based Immunotherapy in the Treatment of FL

DETAILED DESCRIPTION:
Lenalidomide Based Immunotherapy efficacy related molecular biomarker in follicular lymphoma

ELIGIBILITY:
Inclusion Criteria:

Patients diagnose as de novo or relapse refractory FL grade 1-3A .

No history of stem cell transplantation.

Written informed consent.

Exclusion Criteria:

Chemotherapy or large field radiotherapy within 3 weeks prior to entering the study.

Clinically significant active infection.

Impaired liver, renal or other organ function not caused by lymphoma, which will interfere with the treatment schedule.

Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures.

Subject has ≥grade 2 peripheral neuropathy or grade 1 with pain within 14 days before enrollment.

Patients who are pregnant or breast-feeding.

HIV infection.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
CR | 12 weeks
  Complete response rate

SECONDARY OUTCOMES:
PFS | 1 year
  Progression free survival rate
OS | 1 year
  Overall survival rate
ORR | 12 weeks
  Overall response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China